CLINICAL TRIAL: NCT04059133
Title: The Effect of Low Intensity Extracorporeal Low Energy Shock Wave Therapy on Stress Urinary Incontinence and Overactivity Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20180010
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Stress Urinary Incontinence; Overactive Bladder
Keywords: low intensity extracorporeal low energy shock wave therapy; stress urinary incontinence; overactive bladder; urine leakage
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LiESWT arm (Experimental): 1. For SUI: The LiESWT was applied with 0.25 mJ/mm2 intensity, 3000 pulses of shocks, and frequency of 3 pulses/second, once weekly for 4-weeks (W4) and 8-weeks (W8). Probe be transcutaneous applied to the left and right labia minora of the genital area, and the applicator was gently placed on the middle, the left side and the right side of the labia with 0.25 mJ/mm2 intensity and 1000 pulses of shocks individually.
  2. For OAB: The LiESWT was applied with 0.25 mJ/mm2 intensity, 3000 pulses of shocks, and frequency of 3 pulses/second, once weekly for 4-weeks (W4) and 8-weeks (W8). Probe be transcutaneous applied to the lower abdomen with two fingers apart from the pubic symphysis, tilting to 45°, and the applicator was gently placed on suprapubic skin area over the bladder dome and bilateral bladder walls with 0.25 mJ/mm2 intensity and 1000 pulses of shocks individually.
  Interventions: Device: DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL EvoTronTM, GA)-LiESWT arm
- Sham arm (Sham Comparator): 1. For SUI: The LiESWT was applied with 3000 pulses of shocks, frequency of 3 pulses/second but no energy, once weekly for 4-weeks (W4) and 8-weeks (W8). Probe be transcutaneous applied to the left and right labia minora of the genital area, and the applicator was gently placed on the middle, the left side and the right side of the labia with 0.25 mJ/mm2 intensity and 1000 pulses of shocks individually.
  2. For OAB: The LiESWT was applied with 3000 pulses of shocks, frequency of 3 pulses/second but no energy, once weekly for 4-weeks (W4) and 8-weeks (W8). The applicator was gently placed on the suprapubic skin area over the bladder dome (1000 pulses) and bilateral bladder walls (each side 1000 pulses). The probe was placed on the lower abdomen with two fingers apart from the pubic symphysis, tilting to 45°.
  Interventions: Device: DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL EvoTronTM, GA)-Sham arm

INTERVENTIONS:
Device: DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL EvoTronTM, GA)-Sham arm — Sham treatment (shock wave probe w/o energy)
  Arms: Sham arm
Device: DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL EvoTronTM, GA)-LiESWT arm — Low intensity extracorporeal low energy shock wave treatment (shock wave probe w/ energy)
  Arms: LiESWT arm

SUMMARY:
The hypothesis of the present study is low intensity extracorporeal low energy shock wave therapy (LiESWT) can decrease inflammatory disorders, increase pelvic floor blood supply, enhanced bladder stem cell activation, Using LiESWT can decrease bladder overactivity, eliminate urinary incontinence and improve stress urinary incontinence (SUI) and overactive bladder (OAB) symptoms. Therefore improve quality of life and improve social activity.

DETAILED DESCRIPTION:
Clinical application of low intensity extracorporeal low energy shock wave therapy (LiESWT) (2000 to 3000 impulses in 0.20-0.25 millijoule/mm2 (mJ/mm2)) initiated wound healing, promoted angiogenesis, reduced the level of oxidative stress, induced the releasing of VEGF, stimulated proliferation and differentiation of stem cells, and resulted in the effect of anti-inflammatory and tissue regeneration. Generally, LiESWT was used clinically to improve tissue regeneration at tendon-bone junctions, ischemic cardiovascular disorders, skin wound healing, chronic injuries of soft tissues and erectile dysfunction.

LiESWT has also been shown to increase vascular endothelial growth factor (VEGF) expression in ischemic tissues in vivo and to promote angiogenesis and functional recovery in models of chronic myocardial ischemia, myocardial infarction, and peripheral artery disease. Importantly, the advantages of LiESWT include therapies without medication or surgery, outpatient therapies, short treatment sessions, no anesthesia required, and non-invasive therapy.

The hypothesis of the present study is LiESWT can decrease inflammatory disorders, increase pelvic floor blood supply, enhanced bladder stem cell activation, Using LiESWT can decrease bladder overactivity, eliminate urinary incontinence and improve stress urinary incontinence (SUI) and overactive bladder (OAB) symptoms. Therefore improve quality of life and improve social activity.

ELIGIBILITY:
Inclusion Criteria:

1. Women patients within 20~75 years old;
2. OAB symptoms for ≥ 3 months;
3. Frequency of micturition ≥ 8 times daytime as well as 2 times nighttime, and ≥ 2 episodes of urgency per week;
4. Patients have a ≥ 3 month history of experiencing Stress Urinary Incontinence (SUI) per week (self reported);
5. Patients with OAB symptoms including urgency or/and urgency incontinence, urinary frequency and nocturia in the previous 3 months without medical treatments: antimuscarinic or ß3 agonist therapy;
6. Patients can understand, obey order and finish the questionnaires;
7. Patients would like to sign the informed consent;
8. Signature of informed consent form.

Exclusion Criteria:

1. Urinary tract infection (UTI) at screening and recurrent UTI defined as ≥ 3 UTIs in the previous 12 months;
2. Patients who have other disease: diabetes mellitus, spinal cord injury, stoke history, brain disease and neurogenic disease which can cause OAB;
3. Chronic urologic inflammatory condition (Interstitial cystitis, urethral syndrome, painful bladder syndrome);
4. Bladder stone;
5. History of carcinoma of the urinary tract;
6. Lower urinary tract surgery in the last 6 months;
7. Patients who have operation, wound or infection around perineum;
8. Patients who have catheterization due to poor voiding function of urine;
9. Patients who have severe cardiovascular disease;
10. Patients who have severe coagulopathy or liver failure or renal failure;
11. Patients who have underlying urologic cancer;
12. Subjects with gross hematuria;
13. Significant bladder outflow obstruction;
14. Previous pelvic radiation therapy or previous, current malignant disease of the pelvic organs or having received intravesical injection or electrostimulation in the past 12 months;
15. Drug or nondrug treatments of OAB (in the previous 14 days), Concomitant medications that affect detrusor activity;
16. Subjects with history of kidneys stones;
17. Treatable condition that could cause urinary incontinence or urgency;
18. Neurological impairment or psychiatric disorder preventing appropriate understanding of consent and ability to comply with site personnel instructions;
19. History of drug or alcohol abuse within the last 12 months;
20. Within 1 month before entering the test and receive low-energy in vitro shock wave treatment process using antibiotics or phosphodiesterase inhibitors type 5 (PDE5i);
21. There are chronic pelvic pains caused by the merger of other diseases or injuries;
22. Urinary incontinence need to install the catheter;
23. Severe cardiopulmonary disease or diabetes is obviously poor control;
24. Obvious coagulation dysfunction or liver and kidney dysfunction.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Pad Weight Difference | Data will be analyzed at study completion at approximately 3 years.
  The pad test quantifies in grams urinary loss through the absorbent weighing as a measure of stress urinary incontinence.
Overactive bladder symptoms scores (OABSS) | Data will be analyzed at study completion at approximately 3 years.
  Change in OABSS scores during LiESWT treatment and follow-up period.
International Consultation on Incontinence Questionnaire -- Short Form (ICIQ-SF) | Data will be analyzed at study completion at approximately 3 years.
  Change in ICIQ-SF scores during LiESWT treatment and follow-up period.
Urogenital distress inventory (UDI-6) | Data will be analyzed at study completion at approximately 3 years.
  Change in UDI-6 scores during LiESWT treatment and follow-up period.
Incontinence impact questionnaire -7 (IIQ-7) | Data will be analyzed at study completion at approximately 3 years.
  Change in IIQ-7 scores during LiESWT treatment and follow-up period.

SECONDARY OUTCOMES:
maximum flow rate(Qmax=cc/s) | Data will be analyzed at study completion at approximately 3 years.
  The maximum flow rate is the most important uroflowmetry index to diagnose bladder outlet obstruction or bladder contractility.
Uroflow | Data will be analyzed at study completion at approximately 3 years.
  Uroflow curve pattern: There are 5 uroflow curve patterns, bell-shaped, tower-shaped, interrupted-shaped, staccato-shaped and plateau shaped by uroflowmetry. The shape is determined by detrusor contractility and influenced by abdominal straining, coordination with the bladder outlet musculature and any distal anatomic obstruction.
postvoid residual urine volume (PVR) | Data will be analyzed at study completion at approximately 3 years.
  PVR (cc): ultrasonographic bladder scan machines calculates bladder volume. PVR measurements in neurologically intact children are highly variable. PVR must be obtained immediately after voiding(<5min).
3-day micturition diary | Data will be analyzed at study completion at approximately 3 years.
  The mean number of Intake (ml), output (ml), average urine volume (ml), functional bladder capacity (ml), urinary frequency (times/24hrs), urgency (times), and nocturia (times) per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long CY, Lin KL, Lee YC, Chuang SM, Lu JH, Wu BN, Chueh KS, Ker CR, Shen MC, Juan YS. Therapeutic effects of Low intensity extracorporeal low energy shock wave therapy (LiESWT) on stress urinary incontinence. Sci Rep. 2020 Apr 2;10(1):5818. doi: 10.1038/s41598-020-62471-4. PMID 32242035